CLINICAL TRIAL: NCT03670225
Title: Evaluating Clinical Acceptance of a NPWT Wound Care System to Expected Standards of Care in Post-acute Patients With a Variety of Wound Types
Brief Title: Evaluating Clinical Acceptance of a NPWT Wound Care System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medela AG (Industry)
Collaborators: Joseph M. Still Research Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC1801
Record Dates: First submitted 2018-09-07; First posted 2018-09-13 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Foot Ulcer; Pressure Injury; Pressure Ulcer
MeSH Terms: conditions — Diabetic Foot; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Invia Motion Endure (Other)
  Interventions: Device: Invia Motion Endure

INTERVENTIONS:
Device: Invia Motion Endure — NPWT Invia Motion Endure

SUMMARY:
Determine if use of the Medela Invia Motion NPWT system supports acceptable progress towards the goal of therapy when treating patients with a variety of wound types during the evaluation period.

DETAILED DESCRIPTION:
The primary objective of this study is to determine acceptable progress towards the goal of therapy for a diabetic foot ulcers (DFU) and pressure Injuries/ulcers (PI/PU) wounds when using the Medela Invia Motion Endure NPWT system during 4-week study duration.

Goal of therapy will be defined by the physician according to initial assessment:

Endpoints (dependent on goal of therapy):

* Decrease in wound volume
* Decrease in size of the tunneling area
* Decrease in size of undermining
* Decrease in amount of slough
* Increase in granulation tissue
* The wound bed is progressing acceptably towards a transition to another treatment modality such as Moist Wound Healing (MWH), surgical closure, or a flap or graft.

**Study endpoint will be determined by physician at the time of enrollment, when the goal of therapy is documented**

B. Secondary Objectives

* To evaluate the ease of use from clinicians.
* To evaluate overall satisfaction from clinicians. C. Tertiary Objectives
* Adequate management of the exudate

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥18 years of age.
* Signed, informed consent by patient or LAR within 72 hours of admission to burn center.
* Patient is determined to be in need of NPWT for treatment of a diabetic foot ulcer, pressure injuries/pressure ulcer.
* Patient is comfortable (e.g. not in pain)
* Patient is willing and able to adhere to treatment protocol.

Exclusion Criteria:

* Patient not willing to comply with f/u clinic visits.
* Subjects with

  * Necrotic tissue with eschar present
  * Untreated osteomyelitis
  * Non-enteric and unexplored fistulas
  * Malignancy in wound
  * Exposed vasculature
  * Exposed nerves
  * Exposed anastomotic site of blood vessels or bypasses
  * Exposed organs
* Subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
* Patients with concurrent conditions or co-morbidities that in the opinion of the investigator may compromise patient safety or study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Determine if Invia Motion Endure supports acceptable progress towards the goal of therapy for DFU and PI/PU wounds | 4 weeks
  Goal of the therapy will be defined by the physician according to initial assessment:
  * Decrease in wound volume
  * Decrease in size of the tunneling area
  * Decrease in size of undermining
  * Decrease in amount of slough
  * Increase in granulation tissue
  * The wound bed is progressing acceptably towards a transition to another treatment modality such as Moist Wound Healing (MWH), surgical closure, or a flap or graft.
  **Study endpoint will be determined by physician at the time of enrolment, when the goal of therapy is documented**

SECONDARY OUTCOMES:
Evaluation of ease of use and satisfaction | 4 weeks
  A weekly survey will be obtained from the wound clinic staff members to determine ease of use and satisfaction

OTHER OUTCOMES:
Adequate management of the exudate | 4 weeks
  Measurament of exudate (ml, number of canisters used) will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Mullins, MD, Principal Investigator — Joseph M. Still Research Foundation
Locations (1):
- Joseph M. Still Research Foundation, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sen CK, Gordillo GM, Roy S, Kirsner R, Lambert L, Hunt TK, Gottrup F, Gurtner GC, Longaker MT. Human skin wounds: a major and snowballing threat to public health and the economy. Wound Repair Regen. 2009 Nov-Dec;17(6):763-71. doi: 10.1111/j.1524-475X.2009.00543.x. PMID 19903300
- [Background] Morrison Informatics, Inc. A comprehensive cost analysis of medicare home oxygen therapy: A study for the American Association for Homecare. June 27, 2006.
- [Background] C. Marquardt et. al. "Negative pressure wound therapy using PHMB gauze for the management of postoperative subcutaneous surgical site infections" Coloproctology" 36:364-369, 2014